CLINICAL TRIAL: NCT03372395
Title: Lactobacilli Implementation to Restore a Balanced Vaginal Ecosystem: a Promising Solution Against Vaginosis, Vaginitis and HPV Infection
Brief Title: Probiotic Implementation as Help in Solving Vaginal Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Pierluigi Benedetti Panici, Full Professor and Director of Dept Obstetrics and Gynecology, University of Roma La Sapienza
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 3642
Record Dates: First submitted 2017-11-14; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Vaginal Infection; ASC-US
Keywords: probiotics implementation; HPV infection; vaginosis; yeast vaginitis
MeSH Terms: conditions — Vaginitis; Atypical Squamous Cells of the Cervix; Papillomavirus Infections; Vaginal Diseases; Candidiasis, Vulvovaginal

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Standard treatment plus short-term (3 months) vaginal Lactobacillus rhamnosus BMX 54 implementation
  Interventions: Other: Lactobacillus rhamnosus BMX 54
- Group 2 (Experimental): Standard treatment plus long-lasting (6 months) Lactobacillus rhamnosus BMX 54 administration
  Interventions: Other: Lactobacillus rhamnosus BMX 54

INTERVENTIONS:
Other: Lactobacillus rhamnosus BMX 54 — Given once a day for 10 days, once every 3 days for 20 days and then once every 5 days for other 2 months in all patients (probiotics implementation for 3 months comprehensively).

SUMMARY:
Over recent years, a growing interest has developed in microbiota and in the concept of maintaining a special balance between Lactobacillus and other bacteria species in order to promote women's well-being. The aim of the study was to confirm that vaginal Lactobacilli long-lasting implementation in women with HPVinfections and concomitant bacterial vaginosis or vaginitis might be able to help in solving the viral infection, by re-establishing the original eubiosis.

DETAILED DESCRIPTION:
A total of 117 women affected by bacterial vaginosis or vaginitis with concomitant HPV infections were enrolled at Department of Gynecological Obstetrics and Urological Sciences, La Sapienza University, Rome, Italy between February 2015 and March 2016. Women were randomized in two groups, standard treatment (metronidazole 500 mg twice a day for 7 days or fluconazole 150 mg orally once a day for 2 consecutive days) plus short-term (3 months) vaginal Lactobacillus implementation (group 1, short probiotics treatment protocol group, n=60) versus the same standard treatment plus long-lasting (6 months) vaginal Lactobacillus rhamnosus BMX 54 administration (group 2, treatment group, n=57).

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* documented BV or yeast vaginitis associated with HPV-infection documented as PAP-smear abnormalities (ASCUS, L-SIL or H-SIL histologically demonstrated as CIN1) and/or positive for HPV-DNA

Exclusion Criteria:

* pregnancy or breastfeeding
* previous abnormal PAP-smear
* CIN2-3
* concomitant malignancies
* immunological diseases
* severe comorbidities
* prolonged corticosteroid treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of a possible role of probiotics in vaginal infections resolution | 9 months
  Changes in clinical responses (absence of typical symptoms associated with vaginal infections)

SECONDARY OUTCOMES:
Treatment-related adverse events record | 9 months
  Assessed by CTCAE v4.0

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Recine N, Palma E, Domenici L, Giorgini M, Imperiale L, Sassu C, Musella A, Marchetti C, Muzii L, Benedetti Panici P. Restoring vaginal microbiota: biological control of bacterial vaginosis. A prospective case-control study using Lactobacillus rhamnosus BMX 54 as adjuvant treatment against bacterial vaginosis. Arch Gynecol Obstet. 2016 Jan;293(1):101-107. doi: 10.1007/s00404-015-3810-2. Epub 2015 Jul 5. PMID 26142892
- [Derived] Palma E, Recine N, Domenici L, Giorgini M, Pierangeli A, Panici PB. Long-term Lactobacillus rhamnosus BMX 54 application to restore a balanced vaginal ecosystem: a promising solution against HPV-infection. BMC Infect Dis. 2018 Jan 5;18(1):13. doi: 10.1186/s12879-017-2938-z. PMID 29304768